CLINICAL TRIAL: NCT06938958
Title: Characterisation of the Postures Encountered During Surgery and Development of Strategies to Reduce the Risk of Developing Work-related Musculoskeletal Disorders in Surgeons
Brief Title: Ergonomic Challenges for Surgeons; The Problem and Solutions
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: University of Plymouth (Other)
Responsible Party: Sponsor
Other Study IDs: 24WBG122; 350363 (Other: IRAS)
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Musculoskeletal Strain; Ergonomics; Posture
Keywords: Surgeons; Ergonomics; OR; Operating Room; Operating Theatre; Work Related Musculoskeletal Disorders; Strain; Posture; IMU; Computer vision
MeSH Terms: conditions — Sprains and Strains | interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Video and Motion Analysis — 1. Measurements of joint angle, body segment position, static and dynamic postures and posture duration.
  2. Video of Surgeon and Procedure.

SUMMARY:
Work-related musculoskeletal disorders (WMSDs) are highly prevalent among surgeons. Despite growing awareness, there remains a lack of detailed data on the specific postures that contribute to ergonomic risk, particularly within General Surgery. This study aims to characterise postures encountered during open, laparoscopic, and robotic gastrointestinal procedures using wearable sensor technology and video analysis, to inform future ergonomic interventions and training.

A single-centre, prospective observational study of 30 surgical cases will be conducted at University Hospitals Plymouth NHS Trust. Participating surgeons will wear inertial measurement units (IMUs) to record real-time body segment position data whilst performing live surgery. A biomechanical model will then be used to calculate joint angles and whole body posture. Video recordings will be synchronised with IMU data to map posture to surgical tasks. Static and dynamic postures will be analysed using standard ergonomic assessment tools. Alternative tools tailored to surgery will be assessed and proposed. Surgeons will complete questionnaires pre- and post-operatively to report musculoskeletal symptoms. Outcomes will compare ergonomic risk across surgical techniques, identify high-risk procedural steps, and assess the acceptability of wearable technologies in the operating theatre. The data generated will also be used to evaluate, train or refine artificially intelligent camera-based pose estimation models for the operating theatre environment in order to make future ergonomics research and assessment more accessible.

DETAILED DESCRIPTION:
Surgeons often spend long hours in physically demanding positions, which can lead to work-related musculoskeletal disorders (WMSDs) such as neck, shoulder, and back pain. These issues can impact a surgeon's well-being, career longevity, and surgical performance. This study aims to understand the ergonomic challenges surgeons face during major gastrointestinal (GI) surgeries, including open, laparoscopic (keyhole), and robotic procedures. By analysing their posture during operations, researchers hope to develop strategies to reduce the risk of injury.

The study will recruit general surgeons from University Hospitals Plymouth NHS Trust who perform or assist in GI surgeries. Using small motion sensors (Inertial Measurement Units, or IMUs) placed on the surgeons' bodies, researchers will track joint movements, body positions, and posture throughout different surgical techniques. This will help identify which postures and surgical steps are associated with the highest ergonomic risk. Video recordings of surgeries will also be collected to analyse movements and develop future training tools.

Surgeons will complete questionnaires before and after surgery to report any discomfort or pain. The study will compare different surgical techniques to determine which carries the highest risk of injury and which aspects of surgery contribute to poor ergonomics.

By identifying high-risk postures and steps within procedures, this research aims to provide recommendations for ergonomic improvements, such as better training, surgical workstation adjustments, or new tools to help surgeons maintain healthier postures. The results could lead to improved surgeon well-being, safer surgical practices, and longer career sustainability. Findings from this study will be used to develop educational materials and future research in surgical ergonomics.

This study is observational and does not require any changes to standard surgical practice. Both surgeons and patients will provide consent before participation, ensuring ethical research practices.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons performing gastro-intestinal (GI) surgery
* Surgeons assisting GI surgery
* Open, laparoscopic and robotic GI operation
* Informed consent from surgeon
* Informed consent from patient

Exclusion Criteria:

* Pre-existing severe practice-limiting musculoskeletal disorder
* Surgeon not consenting to participation
* Patient not consenting to participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surgeons Performing Major Upper GI Surgery at University Hosptials Plymouth NHS Trust
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Joint angle. | During the operative period, from initial incision to final closure.
  Joint angles (in degrees)
Posture duration. | During the operative period, from incision to closure
  The duration of characterised postures (in minutes)
Posture Variability | During the operative period, from incision to closure
  Angles (in degrees/minute)
Ergonomic Risk | During the operative period, from incision to closure
  RULA Score will be calculated

SECONDARY OUTCOMES:
Compare open, laparoscopic and robotic techniques | During the operative period, from incision to closure
  Joint angles (in degrees)
Compare open, laparoscopic and robotic techniques | During the operative period, from incision to closure
  Postural variability (in degrees/minute)
Identify specific surgical procedures which carry high ergonomic risk | Pre-procedure, immediately post procedure and 24 hours after end of procedure.
  Musculoskeletal symptoms will be assessed pre, intra and post operatively using a self-reported modified Borg CR10 scale symptom questionnaire.
  Sensor and symptom data will be correlated with procedure and technique type.
Create a video library for use in development of educational/training/monitoring tools | During the operative period, from incision to closure
  Video footage of the surgeon will be recorded during the procedure and stored, both for postural assessment during this study and for the creation of a data set that can be used to create a camera vision-based system for further data collection, development of further research and training tools.
Determine the acceptability of sensor-based methods for recording posture data during GI surgery | During the operative period, from incision to closure
  Surgeons will be surveyed regarding their experience of using IMUs for collecting posture data during surgery and this will be used to assess the acceptability of this technology for recording posture data for GI surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Derriford Hospital, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
An anonymised video and motion data library will be shared.